CLINICAL TRIAL: NCT01005147
Title: Effect of Tranexamic Acid on Blood Transfusion in Upper Gastrointestinal Bleeding
Brief Title: Effect of Tranexamic Acid in Upper Gastrointestinal Bleeding
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Gary Kinasewitz, Principal Investigator, University of Oklahoma
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14456
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: tranexamic acid; upper GI bleeding; blood transfusion; GI bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid arm (Experimental)
  Interventions: Drug: tranexamic acid
- Control arm (Placebo Comparator): Will receive a placebo in place of tranexamic acid treatment
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: tranexamic acid — 1 gm every 6 hours for 4 days via IV for non-renal impaired subjects. Alternate IV dosing for renally-impaired subjects: 10mg/Kg BID (1.36 - 2.83 mg/dl clearance); 10mg/Kg QD (2.84 - 5.66 mg/dl clearance; and 10mg/Kg Q48H or 5mg/Kg (.5.66mg/dl clearance)
  Other Names: Cyklokapron
  Arms: Tranexamic acid arm
Other: Placebo — Will receive placebo treatment as per the tranexamic acid schedule
  Arms: Control arm

SUMMARY:
The investigators hypothesize that addition of Tranexamic acid, an antifibrinolytic agent, to conventional therapy will lead to an improved outcome characterized by lower transfusion requirements.

DETAILED DESCRIPTION:
After informed consent is obtained patients will be randomized to receive either Tranexamic acid or placebo in additional to conventional therapy. All patients with gastrointestinal hemorrhage who are admitted to the ICU are managed in consultation with the GI physicians. The ICU team in consultation with the gastroenterology team will manage these patients. Tranexamic acid will be administered in a dose of 1 gm intravenously every 6 hours for four days.

The majority of patients with GI bleeding will spontaneously stop bleeding. However, in those patients that do not and are hemodynamically unstable it poses a significant management challenge. Management of these individuals includes resuscitation followed by endoscopy as well as therapy guided by clinical diagnosis. With optimal therapy mortality in these individuals remains high and the amount of blood transfusion on occasions turns out to be massive and often the outcomes are futile. Tranexamic acid is an antifibrinolytic agent that has been shown to be associated with reduced bleeding and transfusion requirement in surgical patients. We would like to randomize patients to receive either Tranexamic acid or placebo in addition to conventional therapy and monitor outcome.

This study should provide us with information about the efficacy of this medicine in patients with upper GI bleeding. Data from this trial will provide us information about utility of pursuing this modality of therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients with GI bleed if the following criteria are met:

  * has received 4 units of PRBCs within a 24-hour period, or
  * has orthostatic hypotension (drop in SBP of 20mmHg or drop in DBP of 10mmHg after fluid resuscitation with at least 20ml/Kg of either isotonic fluid and/or PRBCs), or
  * if the MAP remains below 60mmHg after fluid resuscitation, and
  * written informed consent is obtained from the subject or legally authorized representative.

Exclusion Criteria:

* Pregnant or lactating women
* Known to have gastrointestinal malignancy
* On anticoagulation therapy
* Patients with history of thromboembolism
* Patients with history of myocardial infarction or ischemic cerebrovascular accident
* Patient with end stage renal disease
* Patients with DNR status
* Incarcerated individuals

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Amount of blood transfusions needed (units of packed RBCs) | Every 6 months

SECONDARY OUTCOMES:
Rebleeding events | Every 6 months
Need for surgical intervention | Every 6 months
Mortality rates | Every 6 months
Length of stay in ICU | Every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jijo John, MD, Principal Investigator — University of Oklahoma; Gary T. Kinasewitz, MD, Principal Investigator — University of Oklahoma